CLINICAL TRIAL: NCT04956484
Title: A Single Arm, 24 Weeks, Pilot Study of Belimumab In Treatment of Early Systemic Lupus Erythematosus
Brief Title: Belimumab In Early Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXM-210622
Record Dates: First submitted 2021-07-08; First posted 2021-07-09 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-04

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: SLE; Belimumab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Belimumab 10 mg/kg plus standard of care (Experimental): Standard of care and Belimumab: 10 mg per kilogram of body weight，days 1 (baseline), 15, and 29 and every 28 days thereafter to week 24
  Interventions: Biological: Belimumab; Drug: Standard of care

INTERVENTIONS:
Biological: Belimumab — Belimumab 10 mg/kg
  Other Names: BENLYSTA™
Drug: Standard of care — Steroid(≤1mg/kg/d) with or without proper immunosuppressants：CTX, MMF, AZA, CsA, FK 506, HCQ, MTX, LEF, SASP etc.

SUMMARY:
To investigate the efficacy of belimumab in early SLE patients (disease duration less than 6 months).

DETAILED DESCRIPTION:
This is a single arm, 24 weeks, pilot trial. All patients will be treated with standard of care plus Belimumab (at a dose of 10 mg per kilogram of body weight) .

The primary endpoint is the proportion of LLDAS in week 24.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE according to the 1997 American College of Rheumatology (ACR) classification criteria or 2019 EULAR/ACR classification criteria within three months, which is autoantibody-positive (antinuclear antibody titers ≥1:80, anti-double-stranded DNA antibodies, or both)
* 18-75 years of age
* body weight 45-80kg
* Disease duration of SLE ≤ 6months
* SELENA-2K score ≥6 scores
* Negative pregnancy test for child-bearing women at screening and baseline
* Provide written informed consent

Exclusion Criteria:

* Known to be allergic to Prednisone Acetate, Meprednisone, Hydroxychloroquine, and Immunosuppressants including Mycophenolate Mofetil, Cyclophosphamide,et al
* Active serious neuropsychiatric systemic lupus erythematosus or other severe situations of SLE who need pulse steroid treatment
* Abnormal liver function (ALT or AST is 2 times higher than normal)
* Pregnancy or breastfeeding women;
* Have a history of malignant tumors;
* Have any serious acute, chronic or recurrent infectious disease (such as pneumonia or active stage of pyelitis, recurrent pneumonia, chronic bronchiectasis and tuberculosis)
* Chronic infections, such as Hepatitis B virus or hepatitis B and C and HIV;
* Previous visual obstruction, monocular dysfunction and cataract;
* Cardiac insufficiency with metabolic imbalance or severe high blood pressure (systolic pressure > 160mmHg or diastolic pressure > 100mmHg) or diabetics;
* Active hemorrhage or peptic ulcer;
* With other concommitant autoimmune disease;
* Receipt of B-cell-targeted therapy (including belimumab) within 1 year before randomization.
* Participated in other drugs clinical trials within 4 weeks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-04-08 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
LLDAS | week 24
  Lupus low disease activity status (LLDAS) was defined as SLEDAI-2K ≤4, no activity in any major organ, no new disease activity feature, PGA ≤1, prednisone ≤7.5 mg/day, and allowance for maintenance of IS and antimalarials

SECONDARY OUTCOMES:
Serologies | week 12, week 24
  Changes in titers of anti-DNA antibody levels
Complement levels | week 12, week 24
  Changes in measures of C3, C4
Dynamics of immune cell subsets | week 12, week 24
  T cell and B cell subsets
Glucocorticoid tapering | week 12, week 24
  A prednisone dose that was decreased≤ 7.5mg/d
Remission | week 12, week 24
  a clinical SLEDAI-2K of 0 (disregarding the serology, including anti-dsDNA and complements), Physician Global Assessment <0.5 (0-3). The patient may be on antimalarials, low-dose glucocorticoids (prednisolone ≤5 mg/day), and/or stable immunosuppressives including biologics
LLDAS | week 12
  Lupus low disease activity status (LLDAS) was defined as SLEDAI-2K ≤4, no activity in any major organ, no new disease activity feature, PGA ≤1, prednisone ≤7.5 mg/day, and allowance for maintenance of IS and antimalarials

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College hospital, Beijing, Dongcheng, China

IPD SHARING:
Plan to Share IPD: No